CLINICAL TRIAL: NCT00661102
Title: A Randomized, Open Label Study Comparing the Efficacy of Topical Corticosteroids or Bepantol in the Prophylaxis of Hand-foot Syndrome in Patients Receiving Oral Xeloda for Treatment of Metastatic Breast Cancer or Colorectal Cancer.
Brief Title: A Study of Prophylactic Treatment for Hand-Foot Syndrome in Patients Treated With Oral Xeloda (Capecitabine).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21419
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Adrenal Cortex Hormones; Capecitabine; Pantothenic Acid

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: capecitabine [Xeloda]; Drug: dexpantenol [Bepantol]
- 2 (Active Comparator)
  Interventions: Drug: Corticosteroids; Drug: capecitabine [Xeloda]
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: Corticosteroids — As prescribed
  Arms: 2
Drug: Placebo — As prescribed
  Arms: 3
Drug: capecitabine [Xeloda] — As prescribed
Drug: dexpantenol [Bepantol] — As prescribed
  Arms: 1

SUMMARY:
This 3 arm study will compare the prophylactic effect of topical corticosteroids, Bepantol or placebo on hand-foot syndrome in patients receiving Xeloda for treatment of metastatic breast cancer, metastatic colorectal cancer or adjuvant treatment of colorectal cancer. Patients who have been receiving oral Xeloda for at least 5 days will be randomized to receive prophylactic treatment with either placebo, topical corticosteroids or Bepantol. The anticipated time on study treatment is until disease progression or development of hand-foot syndrome, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* breast cancer or colorectal cancer patients;
* treated with oral Xeloda for <=5 days;
* lack of hand-foot syndrome (palmar-plantar erythrodysesthesia).

Exclusion Criteria:

* existence of clinical symptoms suggesting hand-foot syndrome;
* use of doxorubicin, 5-FU and/or cytarabine for last 3 months;
* diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2008-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Hand-foot syndrome onset | Event driven
QoL C-30 score | Weeks 7, 13 and 17

SECONDARY OUTCOMES:
Adverse events | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- Brazil (24):
  - Fortaleza, Ceará
  - Salvador, Estado de Bahia
  - Salvador, Bahia, Estado de Bahia
  - Taguatinga, Federal District
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Teresina, Piauí
  - Niterói, Rio de Janeiro
  - Rio de Janeiro, Rio de Janeiro
  - Natal, Rio Grande do Norte
  - Caxias do Sul, Rio Grande do Sul
  - Ijuí, Rio Grande do Sul
  - Lajeado, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Itajaí, Santa Catarina
  - Barretos, São Paulo
  - Campinas, São Paulo
  - Jaú, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - Santos, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo